CLINICAL TRIAL: NCT06948877
Title: "Up-Armoring" At-Risk Military Couples: A Stepped Approach to Early Intervention and Strengthening of Military Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: Family Translational Research Group (Unknown); Texas A&M University (Other); Binghamton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FA8650-17-C-6808
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Couples Therapy; Military Family

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned by in-processing week to the intervention or the control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to a self-directed, online couple intervention offered preventively
  Interventions: Behavioral: ARMOR Online
- Control (No Intervention): Usual resources for relationship assistance in the military

INTERVENTIONS:
Behavioral: ARMOR Online — The online version of ARMOR comprised three core components. The first was an MI-based relationship "check-up" with a brief relationship assessment. In the second component, SMs chose relationship improvement domains from a list of 10 topic areas or modules and watched a short (5-7 minute) video on their chosen area providing (a) evidence-based or evidence-informed psychoeducation, (b) modeling of skills, and (c) practice of the skills. For the third component, SMs were asked MI's "key question" (i.e., "What's the next step?" Miller & Rollnick, 2023) and, if desired, completed a planning module where they were given the opportunity to create a personalized action plan (specifying how they might test any planned changes to see if they had the desired impact).
  Arms: Intervention

SUMMARY:
The study tested whether giving young, partnered military service members access to an online relationship help website would help prevent future relationship problems compared to partnered service member who did not have access to the website

DETAILED DESCRIPTION:
This study tested whether access to a self-directed, online couple intervention offered preventively lessened the occurrence of future negative relationship outcomes (i.e., relationship dysfunction, infidelity, intimate partner violence (IPV) for partnered service members in comparison to the usual resources for relationship assistance in the military. Participants were active-duty military in a committed romantic relationship of at least 6-months duration (N = 581; 37.2% married) who had recently completed basic military training and were transitioning into technical training to learn a specific job skill set. Participants were randomly assigned by in-processing week to the intervention or the control condition. The intervention effect was modeled using both Intent to Treat (ITT) and Complier Average Causal Effect (CACE) approaches.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study, participants had to be: (a) in a committed romantic relationship for at least six months and (b) on active duty (not Guard or Reserve).

Exclusion Criteria:

* Participants with prior military service (i.e., not new to the military who were retraining into a different career field) were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Marital Satisfaction Inventory-Brief (MSI-B; Whisman et al., 2009) | six months
  The MSI-B is a true-false, self-report measure of relationship distress derived from the full The MSI-B is a true-false, self-report measure of relationship distress derived from the full True-false, self-report measure of relationship distress
Family Maltreatment measure (Heyman et al., 2021) | six months
  Whether the participant or partner had engaged in intimate partner violence
Infidelity | six months
  Whether the participant or partner had been intimate with non-partner

CONTACTS AND LOCATIONS:
Locations (1):
- Keesler Air Force Base, Biloxi, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No